CLINICAL TRIAL: NCT02767401
Title: The Success of Opening Single CTO Lesions to Improve Myocardial Viability Study (SOS-comedy)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); First Hospital of China Medical University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2015-22
Record Dates: First submitted 2015-10-18; First posted 2016-05-10 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2018-03

CONDITIONS: Hibernation, Myocardial; Complete Occlusion of Coronary Artery
Keywords: PET-CT; Cardiac magnetic resonance (CMR) imaging; Major adverse cardiac events (MACEs); coronary artery disease
MeSH Terms: conditions — Myocardial Stunning; Cardiovascular Diseases; Coronary Artery Disease | interventions — Stents; Percutaneous Coronary Intervention; Aspirin; Clopidogrel; Ticagrelor; Atorvastatin; Rosuvastatin Calcium; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI using stenting or balloon expansion (Active Comparator): Opening single CTO lesions using drug-eluting stents (such as Xience V and Prime, Endeavor Resolute, Taxus express and Libete, Excel, Partner, BUMA, YINYI, TIVOLI,Firebird2,FireHawk, and Coroflex) or balloon expansion plus optimal medical therapy. Intravascular ultrasound (IVUS),optimal coherence tomgraphy (OCT) or fractional flow reserve (FFR) is used if they are needed. Optimal medical therapy includes dual antiplatelet therapy and statins. And optimal medical therapy should include adequate ventricular rate-limiting medication (i.e. Beta-blocker or rate-limiting calcium antagonist) where appropriate. Anti-angina therapy should be used if the patients have symptoms.
  Interventions: Device: stenting or balloon expansion; Drug: aspirin, clopidogrel, ticagrelor, atorvastatin, rosuvastatin, betaloc
- Optimal medical therapy (No Intervention): Optimal medical therapy. It includes dual antiplatelet therapy and statins. And optimal medical therapy should include adequate ventricular rate-limiting medication (i.e. Beta-blocker or rate-limiting calcium antagonist) where appropriate. Anti-anginal therapy should be used if the patients have symptom.

INTERVENTIONS:
Device: stenting or balloon expansion — all species of drug-eluting stent ((such as Xience, Endeavor, Taxus, Excel, Firebird) implantation or balloon expansion (POBA)
  Other Names: percutaneous coronary intervention
  Arms: PCI using stenting or balloon expansion
Drug: aspirin, clopidogrel, ticagrelor, atorvastatin, rosuvastatin, betaloc — Optimal medical therapy includes dual antiplatelet therapy and statins (aspirin, clopidogrel, ticagrelor, atorvastatin, rosuvastatin, betaloc). And optimal medical therapy should include adequate ventricular rate-limiting medication (i.e. Beta-blocker or rate-limiting calcium antagonist) where appropriate. Anti-anginal therapy should be used if the patients have symptom.
  Arms: PCI using stenting or balloon expansion

SUMMARY:
The purpose of this study is to investigate the effect of percutaneous coronary intervention (PCI) on myocardial viability in coronary artery disease patients with single coronary total occlusion (CTO) lesions.

DETAILED DESCRIPTION:
Patients with coronary artery disease might benefit from successful percutaneous coronary intervention (PCI). However, there is currently no consensus on an optimal treatment modality for single lesions resulting in coronary total occlusion (CTO). Since the other coronary arteries are often lesion-free, or with stenosis of less than 50%, patients often present with no symptoms. Although the expert consensus on CTO lesion suggests reducing the incidence of long-term adverse events via successful revascularization, there are few retrospective studies on single CTO lesions. To date, it is unclear whether successful PCI based on optimal medication treatment (OMT) can increase myocardial viability and the extent of myocardial viability related to prognosis of those CTO patients. Therefore, the aim of this multi-center, prospective, open labeled, non-randomized controlled study was to determine if the improvement to myocardial viability in single CTO patients with successful PCI plus OMT was superior to that of patients with only OMT.

ELIGIBILITY:
Inclusion Criteria:

* History of stable or unstable angina
* LVEF > 35% on transthoracic echocardiography measurement
* Single lesion occluding the coronary artery detected by angiography or MSCTA, with or without stenosis of other coronary arteries (≤ 50% stenotic lesion)
* Availability for follow-up for up to 12 months
* No major barriers to provide written consent

Exclusion Criteria:

* Acute Q-wave myocardial infarction during the latest 3 months
* Revascularization in the non-culprit artery during the latest one month
* Unsuitable for PCI
* Unable to tolerate dual antiplatelet treatment (DAPT)
* Severe abnormal hematopoietic system, such as platelet count of < 100×109/L or > 700×109/L and white blood cell count of < 3×109/L
* Active bleeding or bleeding tendency
* Severe coexisting conditions, such as severe renal insufficiency (GFR < 60 ml/min•1.73m2), severe hepatic dysfunction [elevated ALT (glutamic-pyruvic transaminase) or AST (glutamic-oxal acetic transaminase) level by more than three-fold of the normal limitation], acute or chronic heart failure (NYHA III-IV), acute infectious diseases, immune disorders, malignancy, etc.
* Life expectancy < 12 months
* Pregnancy or planning pregnancy
* Drug allergies or contraindications to aspirin, clopidogrel, ticagrelor, statins, contract, anticoagulant, stent, etc.
* Participation or planning to participate in another clinical trial during the same period
* Refusal to comply with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Changes to myocardial viability | 12 months
  Changes to myocardial viability from baseline assessed with the use of combined positron emission tomography and computerized tomography (PET-CT) system

SECONDARY OUTCOMES:
Major adverse cardiac events | 12 months
  including all-cause mortality, cardiac death, first or recurrent acute myocardial infarction, recurrent angina, target lesion revascularization (TLR), heart failure, and re-hospitalization
The rates of target vascular revascularization (TVR), TLR, and stent thrombosis | 12 months
Changes to left ventricular ejection fraction (LVEF) | 12 months
  Changes to LVEF in % assessed with the use of cardiac MRI and transthoracic echocardiography (TTE).
Changes to myocardial infarct size | 12 months
  Changes to myocardial infarct size in percentage of total myocardial size assessed with the use of cardiac MRI.
Changes to left ventricular mass (LVM) | 12 months
  Changes to LVM in g assessed with the use of cardiac MRI.
Changes to cardiac output (CO) | 12 months
  Changes to cardiac CO in in L/min/m2 assessed with the use of cardiac MRI.
Changes to stroke volume (SV) | 12 months
  Changes to SV in ml assessed with the use of cardiac MRI.
Changes to maximum left ventricular ejection rate | 12 months
  Changes to maximum left ventricular ejection rate in % assessed with the use of cardiac MRI.
Changes to maximum left ventricular filling rate | 12 months
  Changes to maximum left ventricular filling rate in % assessed with the use of cardiac MRI.
Changes to maximum slope | 12 months
  Changes to maximum slope assessed with the use of cardiac MRI.
Changes to left ventricular end-diastolic diameter (LVEDd) | 12 months
  Changes to LVEDd in mm assessed with the use of TTE.
Changes to left ventricular end-systolic diameter (LVESd) | 12 months
  Changes to LVESd in mm assessed with the use of TTE.
Changes to cardiac systolic function | 12 months
  Changes to cardiac systolic function in E/A, E'/A', Ea/Aa, EDT in ms assessed with the use of TTE.

OTHER OUTCOMES:
Stroke incidence | 12 months
The number of compliant patients | 12 months
  Compliant patients are usually defined as those who take predefined percentage (100%) of the treatment
The total cost of medical care | 12 months
  The total cost of medical care include equipment and medication in dollars.
Number of guidewires | 12 months
  Number of guidewires used in the procedure
Number of balloons | 12 months
  Number of balloons used in the procedure
Number of stents | 12 months
  Number of stents used in the procedure
the volume of contrast | 12 months
  the volume of contrast in ml during the procedure
type of device | 12 months
  type of the first guidewire and the final guidewire to cross the proximal lesion such as shaping ribbon or core-to-tip, coil or polymer Cover, hydrophilic coating or hydrophobic coating, and the new devices including Guidezilla™， CrossBoss™ , Tornus, Transporter and Stingray™, any other newest device which will be used before this study is completed.
the composite number of special techniques used in the procedure | 12 months
  the special techniques including parallel wire, see-saw technique, side branch technique, STAR (subintimal tracking and reentry), intravascular ultrasound guiding wire, reverse-controlled antegrade and retrograde subintimal tracking (CART) technique and reverse CART technique.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, M.D., Principal Investigator — The First Affiliated Hospital of Dalian Medical University

REFERENCES:
- [Background] Namazi M, Safi M, Vakili H, Saadat H, Alipour S, Mahjoob P, Taherkhani M, Pedari S, Taherion M, Rajabi Moghaddam H, Alhazifi A, Vatanparast M, Khaligh S. Evaluation of effective factors in success rate of intervention on CTO. Acta Med Iran. 2015;53(3):173-6. PMID 25796024
- [Background] Stuijfzand WJ, Raijmakers PG, Driessen RS, van Royen N, Nap A, van Rossum AC, Knaapen P. Value of Hybrid Imaging with PET/CT to Guide Percutaneous Revascularization of Chronic Total Coronary Occlusion. Curr Cardiovasc Imaging Rep. 2015;8(7):26. doi: 10.1007/s12410-015-9340-2. PMID 26029338
- [Background] Lee SH, Yang JH, Choi SH, Song YB, Hahn JY, Choi JH, Kim WS, Lee YT, Gwon HC. Long-Term Clinical Outcomes of Medical Therapy for Coronary Chronic Total Occlusions in Elderly Patients (>/=75 Years). Circ J. 2015;79(8):1780-6. doi: 10.1253/circj.CJ-15-0041. Epub 2015 May 28. PMID 26017064